CLINICAL TRIAL: NCT06736041
Title: A Phase 3, Randomized, Modified Double-blind, Active-controlled, Parallel-group, 2-arm Study to Investigate the Safety and Immunogenicity of a 4-dose Regimen of a 21-valent Pneumococcal Conjugate Vaccine in Healthy Infants and Toddlers
Brief Title: Study of a 4-Dose Regimen of a 21-valent Pneumococcal Conjugate Vaccine in Healthy Infants From Approximately 2 Months of Age
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PSK03; U1111-1294-7860 (Other: WHO ICTRP)
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Pneumococcal Immunization
MeSH Terms: interventions — RotaTeq; Vaxelis; Chickenpox Vaccine; DTaP-IPV-HB-PRP-T vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Modified double-blind
  * Blinding for vaccine group assignment: participants and participant's parent(s) / legally acceptable representative(s) (LARs), outcome assessors, Investigators, laboratory personnel, and Sponsor study staff
  * No blinding for vaccine group assignment: those preparing and administering the study interventions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: PCV21 (Experimental): Participants will be administered via intramuscular injection (IM) a 3-dose primary series of PCV21 at approximately 2, 4 and 6 months of age (MoA) co- administered with Vaxelis or Hexaxim (for participants included in South Korea only) and RotaTeq. At toddler age (12 to 15 MoA), a 4th dose of PCV21 will be administered concomitantly with a single dose of M-M-M-R II and Varivax.
  Interventions: Biological: PCV21 vaccine; Biological: M-M-R II vaccine; Biological: RotaTeq; Biological: Vaxelis vaccine; Biological: Varivax; Biological: Hexaxim Vaccine
- Group 2: 20vPCV (Active Comparator): Participants will be administered via intramuscular injection (IM) a 3-dose primary series of 20vPCV at approximately 2, 4 and 6 months of age (MoA) co- administered with Vaxelis or Hexaxim (for participants included in South Korea only) and RotaTeq. At toddler age (12 to 15 MoA), a 4th dose of 20vPCV will be administered concomitantly with a single dose of M-M-M-R II and Varivax.
  Interventions: Biological: Prevnar 20 vaccine; Biological: M-M-R II vaccine; Biological: RotaTeq; Biological: Vaxelis vaccine; Biological: Varivax; Biological: Hexaxim Vaccine

INTERVENTIONS:
Biological: PCV21 vaccine — Pharmaceutical form:Suspension for injection-Route of administration:Intramuscular
  Other Names: 515
  Arms: Group 1: PCV21
Biological: Prevnar 20 vaccine — Pharmaceutical form:Suspension for injection-Route of administration:Intramuscular
  Other Names: Prevnar20®
  Arms: Group 2: 20vPCV
Biological: M-M-R II vaccine — Pharmaceutical form:Powder, lyophilized, for suspension for reconstitution-Route of administration:Subcutaneous or Intramuscular
  Other Names: M-M-R® II
Biological: RotaTeq — Pharmaceutical form:Solution-Route of administration:Oral
  Other Names: RotaTeq®
Biological: Vaxelis vaccine — Pharmaceutical form:Suspension for injection-Route of administration:Intramuscular
  Other Names: Vaxelis®
Biological: Varivax — Pharmaceutical form:Powder, lyophilized, for suspension for reconstitution-Route of administration:Subcutaneous or Intramuscular
  Other Names: Varivax®
Biological: Hexaxim Vaccine — Pharmaceutical form:Suspension for injection-Route of administration:Intramuscular
  Other Names: Hexaxim®

SUMMARY:
This study is a Phase 3, randomized, modified double-blind study which aims to measure whether PCV21 vaccine (investigational pneumococcal conjugate vaccine) is safe and can help the body to develop germ-fighting agents called "antibodies" (immunogenicity) compared with 20-valent pneumococcal vaccine (Prevnar 20, licensed pneumococcal conjugate vaccine) when they are administered with routine pediatric vaccines in infants aged from approximately 2 months (42 to 89 days).

The study duration per participant will be up to approximately 19 months. The study vaccines (either PCV21 or 20-valent pneumococcal vaccines) will be administered at approximately 2, 4, 6 and 12 to 15 months of age. Routine pediatric vaccines will be given at the same timepoints.

There will be 6 study visits:

-Visit (V)01, V02 separated from V01 by 60 days, V03 separated from V02 by 60 days, V04 separated from V03 by 30 days, V05 at 12 months of age until 15 months of age, V06 separated from V05 by 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Aged 42 to 89 days on the day of inclusion
* Participants who are healthy as determined by medical evaluation including medical history and physical examination
* Born at full term of pregnancy (≥ 37 weeks) and with a birth weight ≥ 2.5 kg or born after a gestation period above 28 (> 28 weeks) through 36 weeks with a birth weight ≥ 1.5 kg, and in both cases medically stable as assessed by the investigator

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy; or long-term systemic corticosteroid therapy
* History of microbiologically confirmed Streptococcus pneumoniae infection or disease
* Any contraindication to the routine pediatric vaccines being administered in the study
* History of seizure or significant stable or progressive neurological disorders such as infantile spasms, inflammatory nervous system diseases, encephalopathy, cerebral palsy
* Known systemic hypersensitivity to any of the study interventions components, or history of a life-threatening reaction to the study interventions used in the study or to a product containing any of the same substances
* Laboratory-confirmed or known thrombocytopenia, as reported by the parent/legally acceptable representative (LAR), contraindicating intramuscular (IM) injection
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM injection
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with study conduct or completion
* Moderate or severe acute illness/infection (according to investigator judgment) or febrile illness (temperature ≥ 38.0°C [≥ 100.4°F]) on the day of study intervention administration. A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
* Receipt of any vaccine in the 4 weeks preceding the study intervention administration or planned receipt of any vaccine in the 4 weeks following the study intervention administration, except for US licensed influenza vaccination, which may be received at least 2 weeks before or 2 weeks after any study vaccination. This exception includes monovalent pandemic influenza vaccines and multivalent influenza vaccines, as applicable per local recommendations.
* Previous vaccination against S. pneumoniae
* Previous vaccination against the following antigens: diphtheria, tetanus, pertussis, Haemophilus influenzae type b, and poliovirus
* Receipt of more than 1 dose of hepatitis B vaccine
* Receipt of immune globulins, blood or blood-derived products since birth
* Participation at the time of study enrollment (or in the 6 weeks preceding the first study intervention administration) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure

Note: The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Ages: 42 Days to 89 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1630 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2027-05-17 (Estimated); Study Completion 2027-05-17 (Estimated)

PRIMARY OUTCOMES:
Seroresponse rate for PCV21 serotypes | 30 days post-dose 3
  Serotype specific IgG concentration ≥ 0.35 µg/mL
IgG concentration for PCV21 serotypes | 30 days post-dose 3
  Serotype specific IgG Geometric Mean Concentration (GMC)
IgG concentration for PCV21 serotypes | 30 days post-dose 4
  Serotype specific IgG GMC post-dose 4

SECONDARY OUTCOMES:
Anti- hepatitis B surface antigen (HBsAg) Ab | 30 days post-dose 3
  % Antibody concentrations ≥ 10 milli international units per milliliter (mIU/mL)
Anti- polyribosylribitol phosphate (PRP) Ab | 30 days post-dose 3
  % Antibody concentrations ≥ 0.15 micrograms per milliliter (µg/mL)
Anti-poliovirus types (1, 2, and 3) Ab | 30 days post-dose 3
  % Antibody titers ≥ 1:8
Anti-diphtheria Ab concentrations | 30 days post-dose 3
  % Antibody concentrations ≥ 0.1 IU/mL
Anti-tetanus Ab concentrations | 30 days post-dose 3
  % Antibody concentrations ≥ 0.1 IU/mL
Anti-pertussis Ab concentrations (Pertussis toxin (PT) and Filamentous Hemagglutinin (FHA)) | 30 days post-dose 3
  Antibody GMC
Anti-rotavirus serum immunoglobulin A (IgA) Ab concentrations | 30 days post-dose 3
  Antibody GMC
Anti-measles Ab concentrations | 30 days post-dose 4
  % Antibody concentrations ≥ 225 milli international units per milliliter (mIU/mL)
Anti-measles Ab concentrations | 30 days post-dose 4
  Antibody GMC
Anti-mumps Ab concentrations | 30 days post-dose 4
  % Anti-mumps Ab concentrations ≥ 10 Ab units (AbU)/mL
Anti-mumps Ab concentrations | 30 days post-dose 4
  Antibody GMC
Anti-rubella Ab concentrations | 30 days post-dose 4
  % Anti-rubella Ab concentrations ≥ 10 IU/mL
Anti-rubella Ab concentrations | 30 days post-dose 4
  Antibody GMC
Anti-varicella Ab concentrations | 30 days post-dose 4
  Anti-varicella Ab concentrations ≥ 5 glycoprotein enzyme linked immunosorbent assay (gpELISA) units/mL
IgG concentration for the additional serotype 9N | 30 days post-dose 3
  Serotype 9N specific IgG concentration ≥ 0.35 µg/mL
IgG concentration for serotype 3 | 30 days post-dose 3
  Serotype 3 specific IgG concentration ≥ 0.35 µg/mL
IgG concentration for additional serotype 9N | 30 days post-dose 3
  Serotype 9N specific IgG GMC
IgG concentration for serotype 3 | 30 days post-dose 3
  Serotype 3 specific IgG GMC
Serotype 9N specific IgG GMC post-dose 4 | 30 days post-dose 4
  Serotype 9N specific IgG GMC post-dose 4
IgG concentration for additional serotype 9N | 30 days post-dose 4
  Serotype 9N specific IgG GMC post-dose 4
IgG concentration for serotype 3 | 30 days post-dose 4
  Serotype 3 specific IgG GMC post-dose 4
Seroresponse rate for PCV21 serotypes | 30 days post-dose 4
  Serotype specific IgG concentration ≥ 0.35 µg/mL
IgG concentration for PCV21 serotypes | Before dose 4 and 30 days post-dose 4
  Serotype specific IgG GMC prior to and post-dose 4
Serotype specific OPA titers for all serotypes included in PCV21 | 30 days post-dose 3
  Antibody GMC
Serotype specific OPA titers ≥ lower limit of quantitation (LLOQ) for all serotypes included in PCV21 | 30 days post-dose 3
  Antibody GMC
Serotype specific OPA titers for all serotypes included in PCV21 | Before dose 4 and 30 days post-dose 4
  Antibody GMC prior to and post-dose 4
Serotype specific OPA titers ≥ lower limit of quantitation (LLOQ) for all serotypes included in PCV21 | Before dose 4 and 30 days post-dose 4
  Antibody GMC prior to and post-dose 4
Presence of any immediate adverse events (AEs) | Within 30 minutes after each vaccine injection
  Number of participants experiencing solicited and unsolicited immediate AEs
Presence of solicited injection site and systemic reactions through 7 days after each vaccine injection | Through 7 days after each vaccine injection
  Number of participants experiencing solicited injection site and systemic reactions
Presence of unsolicited (spontaneously reported) injection site reactions and unsolicited systemic AEs through 30 days after each vaccine injection | Through 30 days after each vaccine injection
  Number of participants experiencing unsolicited injection site reactions and unsolicited systemic AEs
Presence of serious adverse events (SAEs) throughout the study (through 6 months post- last vaccine injection) | Throughout the study (through 6 months post-last vaccine injection), approximately 20 months
  Number of participants experiencing SAEs

CONTACTS AND LOCATIONS:
Locations (103):
- United States (57):
  - Sun City Clinical Research- Site Number : 8400247, Glendale, Arizona
  - Eclipse Clinical Research- Site Number : 8400029, Tucson, Arizona
  - Northwest Arkansas Pediatric Clinic- Site Number : 8400030, Fayetteville, Arkansas
  - Southland Clinical Research Center- Site Number : 8400243, Fountain Valley, California
  - Century Research Institute- Site Number : 8400065, Huntington Park, California
  - Matrix Clinical Research - Huntington Park- Site Number : 8400012, Huntington Park, California
  - Matrix Clinical Research - Los Angeles- Site Number : 8400013, Los Angeles, California
  - FOMAT Medical Research - Pediatric, Infant & Adolescence Medicine- Site Number : 8400063, Ventura, California
  - Velocity Clinical Research - Washington DC- Site Number : 8400049, Washington D.C., District of Columbia
  - PAS Research- Site Number : 8400123, Clearwater, Florida
  - Prohealth Research Center- Site Number : 8400159, Doral, Florida
  - NurtureGen Research- Site Number : 8400205, Homestead, Florida
  - Dade Research Center- Site Number : 8400007, Miami, Florida
  - EMDA Clinical Research- Site Number : 8400237, Miami, Florida
  - Acevedo Clinical Research Associates- Site Number : 8400089, Miami, Florida
  - Miami Clinical Research Tower- Site Number : 8400189, Miami, Florida
  - Bio-Medical Research- Site Number : 8400147, Miami, Florida
  - High Quality Research- Site Number : 8400245, Miami, Florida
  - Riveldi Biomedical Research and Associates - Miami Lakes- Site Number : 8400032, Miami Lakes, Florida
  - BioResearch Partner (BRP) - Premium Healthcare Medical Center - Miami Lakes- Site Number : 8400203, Miami Lakes, Florida
  - Optimal Research Sites- Site Number : 8400232, Orange City, Florida
  - SEC Clinical Research - Pensacola- Site Number : 8400003, Pensacola, Florida
  - National Clinical Trials - Tampa- Site Number : 8400229, Tampa, Florida
  - PAS Research - Tampa- Site Number : 8400002, Tampa, Florida
  - Medical Research Partners - Ammon- Site Number : 8400239, Ammon, Idaho
  - Bingham Memorial Hospital - Blackfoot- Site Number : 8400084, Blackfoot, Idaho
  - Leavitt Women's Healthcare- Site Number : 8400085, Idaho Falls, Idaho
  - Snake River Research- Site Number : 8400060, Idaho Falls, Idaho
  - Clinical Research Prime Rexburg- Site Number : 8400250, Rexburg, Idaho
  - Alliance for Multispeciality Research - El Dorado- Site Number : 8400010, El Dorado, Kansas
  - Hutchinson Clinic- Site Number : 8400061, Hutchinson, Kansas
  - Cotton O'Neil Pediatrics- Site Number : 8400009, Topeka, Kansas
  - KUR Research at Columbia MD - 6220 Old Dobbin Lane- Site Number : 8400242, Columbia, Maryland
  - Michigan Institute of Research- Site Number : 8400207, Allen Park, Michigan
  - University of Missouri Hospital- Site Number : 8400244, Columbia, Missouri
  - Vector Clinical Trials- Site Number : 8400249, Las Vegas, Nevada
  - Prime Global Research- Site Number : 8400246, The Bronx, New York
  - Monroe Biomedical Research - Monroe- Site Number : 8400225, Monroe, North Carolina
  - Dayton Clinical Research- Site Number : 8400087, Dayton, Ohio
  - Allegheny Health Network - Health and Wellness Pavilion- Site Number : 8400111, Erie, Pennsylvania
  - Tribe Clinical Research - Greenville - Verdae Boulevard- Site Number : 8400005, Greenville, South Carolina
  - Coastal Carolina Research Center - North Charleston- Site Number : 8400064, North Charleston, South Carolina
  - Inquest Clinical Research - Baytown - West Baker Road- Site Number : 8400112, Baytown, Texas
  - South Texas Clinical Research- Site Number : 8400025, Corpus Christi, Texas
  - FamilyHealthWatch - KeyPoint Clinical Research- Site Number : 8400173, Dallas, Texas
  - Helios Clinical Research - Fort Worth - 8th Avenue- Site Number : 8400072, Fort Worth, Texas
  - Ventavia Research Group - Houston - North Loop West- Site Number : 8400093, Houston, Texas
  - Gonzalez Family & Occupational Medicine- Site Number : 8400035, Houston, Texas
  - La Providence Pediatrics & Family Clinics- Site Number : 8400026, Houston, Texas
  - Houston Clinical Research Associates- Site Number : 8400018, Houston, Texas
  - LinQ Research, LLC - Katy- Site Number : 8400258, Katy, Texas
  - Maximos Ob/Gyn- Site Number : 8400056, League City, Texas
  - Pediatric Center - Richmond- Site Number : 8400068, Richmond, Texas
  - Tanner Clinic- Site Number : 8400241, Layton, Utah
  - Wasatch Pedicatrics- Site Number : 8400153, Murray, Utah
  - Rio Clinical Trials - Canyon View- Site Number : 8400222, Ogden, Utah
  - Clinical Research Partners - Richmond - Forest Avenue- Site Number : 8400236, Richmond, Virginia
- Australia (5):
  - Investigational Site Number : 0360001, Westmead, New South Wales
  - Investigational Site Number : 0360004, Brisbane, Queensland
  - Investigational Site Number : 0360005, Southport, Queensland
  - Investigational Site Number : 0360002, Parkville, Victoria
  - Investigational Site Number : 0360003, Perth, Western Australia
- Honduras (3):
  - Investigational Site Number : 3400001, San Pedro Sula
  - Investigational Site Number : 3400002, Tegucigalpa
  - Investigational Site Number : 3400003, Tegucigalpa
- Puerto Rico (6):
  - Investigational Site Number : 6300004, Caguas
  - Investigational Site Number : 6300008, Guayama
  - Investigational Site Number : 6300003, Ponce
  - Investigational Site Number : 6300002, San Juan
  - Investigational Site Number : 6300006, San Juan
  - Investigational Site Number : 6300005, Trujillo Alto
- South Korea (29):
  - Investigational Site Number : 4100023, Busan, Busan
  - Investigational Site Number : 4100030, Daegu, Daegu
  - Investigational Site Number : 4100024, Daegu, Daegu
  - Investigational Site Number : 4100034, Gwangju, Gwangju
  - Investigational Site Number : 4100020, Ansan-si, Gyeonggi-do
  - Investigational Site Number : 4100002, Anyang-si, Gyeonggi-do
  - Investigational Site Number : 4100013, Bucheon-si, Gyeonggi-do
  - Investigational Site Number : 4100029, Bucheon-si, Gyeonggi-do
  - Investigational Site Number : 4100014, Hwaseong-si, Gyeonggi-do
  - Investigational Site Number : 4100011, Seongnam-si, Gyeonggi-do
  - Investigational Site Number : 4100001, Seongnam-si, Gyeonggi-do
  - Investigational Site Number : 4100027, Changwon-si, Gyeongsangnam-do
  - Investigational Site Number : 4100010, Yangsan, Gyeongsangnam-do
  - Investigational Site Number : 4100017, Bupyeong-gu, Incheon-gwangyeoksi
  - Investigational Site Number : 4100006, Incheon, Incheon-gwangyeoksi
  - Investigational Site Number : 4100025, Jeonju, Jeollabuk-do
  - Investigational Site Number : 4100019, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100008, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100005, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100004, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100009, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100015, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100007, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100031, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100003, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100026, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100022, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100018, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100016, Seoul, Seoul-teukbyeolsi
- Thailand (3):
  - Investigational Site Number : 7640007, Bangkok
  - Investigational Site Number : 7640005, Bangkok
  - Investigational Site Number : 7640004, Khon Kaen

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Pichon S, Ullery GM, Cousin L, Sadarangani M, Ryu JH, Monfredo C, Mari K, Pandey A, Personnic S, Pouzet C, Manson C, Silhadi W, Minutello AM. Safety and Immunogenicity of a Pneumococcal Conjugate Vaccine When Administered Concomitantly With Routine Pediatric Vaccines in Healthy Toddlers and Infants. Pediatr Infect Dis J. 2025 Oct 1;44(10):995-1008. doi: 10.1097/INF.0000000000004913. Epub 2025 Jul 31. PMID 40833801
- See also: PSK03 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26364&tenant=MT_SNY_9011